CLINICAL TRIAL: NCT03502356
Title: ADDATION OF Azithromycin TO CEFAZOLIN PRE ELECTIVE C S
Brief Title: Addition of Azithromycin to Cefazolin Will Reduce Post CS Infections More Than Cefazolin Only.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mohamed abd elhamied abd elgaber, cario egypt, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2377
Record Dates: First submitted 2018-04-11; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Randomized Controll Trial
MeSH Terms: interventions — Azithromycin; Cefazolin

STUDY DESIGN:
Intervention Model Description: Control Group:
  This group will include 200women undergoing elective cs. In this group, patients will receive standard antibiotic prophylaxis CEFAZOLIN (at a dose of 1 g) and azithromycin (at a dose of 1g) 2 hours preoperative.
  Study Group:
  This group will include 200women undergoing elective cs. In this group, patients will receive only standard prophylaxis antibiotic(CEFAZOLIN)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): This group will include 200women undergoing elective cs. In this group, patients will receive standard antibiotic prophylaxis CEFAZOLIN (at a dose of 1 g) and azithromycin (at a dose of 1g) 2 hours preoperative.
  Interventions: Drug: Azithromycin
- Study Group (No Intervention): This group will include 200women undergoing elective cs. In this group, patients will receive only standard prophylaxis antibiotic(CEFAZOLIN)

INTERVENTIONS:
Drug: Azithromycin — In this group, patients will receive standard antibiotic prophylaxis CEFAZOLIN (at a dose of 1 g) and azithromycin (at a dose of 1g) 2 hours preoperative.
  Other Names: Cefazolin
  Arms: Control Group

SUMMARY:
The good standard antibiotic prophylaxis pre elective C S is cefazolin and this study will approve addition of azithromycin to cefazolin will reduce post CS infections more than cefazolin only.

DETAILED DESCRIPTION:
Patiants and methods

Randomization:

Patients fulfilling the inclusion criteria will be randomized to two groups. Both two group will receive standard prophylaxis antibiotic CEFAZOLIN (zinol) (at a dose of 1 g) 2 hours preoperative.

Control Group:

This group will include 200women undergoing elective cs. In this group, patients will receive standard antibiotic prophylaxis CEFAZOLIN (at a dose of 1 g) and azithromycin (at a dose of 1g) 2 hours preoperative.

Study Group:

This group will include 200women undergoing elective cs. In this group, patients will receive only standard prophylaxis antibiotic(CEFAZOLIN)

Inclusion criteria:

* Gestational age of 37 0/7 weeks and greater
* Elective cesarean section
* Medicaly free pregnant women

Exclusion criteria:

* a known allergy to azithromycin
* obstetric complications
* azithromycin use within 7 days before randomization
* chorioamnionitis or other infection requiring postpartum antibiotic therapy
* Pre-gestational diabetes

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 37 0/7 weeks and greater
* Elective cesarean section
* Medicaly free pregnant women

Exclusion Criteria:

* a known allergy to azithromycin
* obstetric complications
* azithromycin use within 7 days before randomization
* chorioamnionitis or other infection requiring postpartum antibiotic therapy
* Pre-gestational diabetes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-04-20 (Estimated); Primary Completion 2018-06-20 (Estimated); Study Completion 2018-08-20 (Estimated)

PRIMARY OUTCOMES:
endometritis | 6 weeks after surgery
  Endometritis was defined as the presence of at least two of the following signs with no other recognized cause: fever (temperature of at least 38°C [100.4°F]), abdominal pain, uterine tenderness, or purulent drainage from the uterus

CONTACTS AND LOCATIONS:
Overall Officials: mohamed 20 amar, md, Study Chair — ain shams
Locations (1):
- Ain Shams, Cairo, Elabasy, Egypt